CLINICAL TRIAL: NCT05297227
Title: Non-surgical Periodontal Therapy: Efficacy of Repeated Subgingival Instrumentation for Non-responding Sites. A Quasi-experimental Study
Brief Title: Non-surgical Periodontal Therapy: Efficacy of re Treatment for Non-responding Sites.
Acronym: Nrs_1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Associate Professor, University of Siena
Other Study IDs: Nrs_1
Record Dates: First submitted 2022-03-16; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Periodontal Therapy; Non Responding Sites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Non surgical periodontal Therapy — Non-surgical periodontal therapy comprising oral hygiene instruction and motivation, professional mechanical plaque removal, and subgingival instrumentation will be performed. It consists in the use of an ultrasuond (piezoeletric device) and manual curettes.

SUMMARY:
The current experimental protocol is a pre-post quasi-experimental design. A cohort of individuals will be enrolled progressively according to a screening record of periodontitis. They were treated with PMPR and Subgingival Instrumentation according to their diagnosis. After 3 months they will be re-evaluated, and non-responding sites (Ppd>=4mm and bop+) will be scheduled for the second session of PMPR and SI. After 2 months they will be re-evaluated and clinical efficacy will be defined.

DETAILED DESCRIPTION:
The current experimental protocol is a pre-post quasi-experimental design. A cohort of individuals will be enrolled progressively according to a screening record of periodontitis. Once included, individuals will receive, by a calibrated examiner, a full-mouth periodontal chart, and accordingly, they will be treated in a multi-step approach, in accordance with the recent clinical guidelines. The treatment will consist of oral hygiene instruction and motivation, risk factor control, professional mechanical plaque removal (PMPR), and subgingival instrumentation (SI): it will be performed by two experienced operators. Thereafter, after 3 months, patients will be evaluated and a new periodontal chart will be performed. The presence of non-responding sites (Ppd>4 and bop+) will be treated with the second session of PMPR plus Subgingival Instrumentation. After 2 months patients will be clinically evaluated and a full periodontal chart will be completed.

ELIGIBILITY:
Inclusion Criteria:

* unremarkable general health; age 18-80; minimum of 20 teeth; Periodontitis (Stage 1-4); no antibiotic intake in the previous 6 months;

Exclusion Criteria:

* Subgingival instrumentation in the previous 12 months
* No antibiotic intake in the previous 3 months
* A compromised medical condition requiring prophylactic antibiotic coverage
* Pregnant/nursing
* Ongoing drug therapy that might alter the clinical signs and symptoms of periodontitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with a Diagnosis of Periodontitis were recruited consecutively after a full mouth clinical examination and radiographic evaluation. The screening and periodontal chart were performed at the Department of Medical Biotechnologies, Unit of Periodontology, University Hospital of Siena, Siena (Italy).
Sampling Method: Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of pocket closures | through study completition, 6 months
  Proportion of pathological periodontal pockets (non responding site) that will be closed (Ppd <5 and bop-) after the second instrumentation